CLINICAL TRIAL: NCT04331210
Title: Rectal Versus Oral Diclofenac Sodium in Relieving Post Episiotomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hosny Ahmed, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Post episiotomy analgesia
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Episiotomy Wound
Keywords: Episiotomy
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Using diclofenac sodium suppository 50 mg immediately after suturing and then every 8 hours
  Interventions: Drug: Diclofenac Sodium
- Group 2 (Active Comparator): Using diclofenac sodium tablets 50 mg every 8 hours after birth
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Diclofenac Sodium — Group 1 will take oral diclofenac sodium and group 2 will take Rectal diclofenac sodium as an analgesic

SUMMARY:
Current study aims to compare oral diclofenac sodium with it's rectal form for analgesia of pain after episiotomy.

DETAILED DESCRIPTION:
* Episiotomy is a surgical incision of the perineum and the posterior vaginal wall.
* it can be done at a 60 degree angle from the vulva towards the anus or at an angle from the posterior end of the vulva.
* usually under local anesthetic and is sutured after delivery.
* It is done during second stage of labor to enlarge the opening for the baby to pass through to avoid soft-tissue tearing which may involve the anal sphincter and rectum.
* Perineal pain after episiotomy has immediate and long-term negative effects for women and their babies. These effects can interfere with breastfeeding and the care of the infant.
* Usually women undergo episiotomy need a good analgesic to overcome pain resulting from the analgesic.
* Previous study by Faiza shafi, Shazia sayed, Naheed bano, Rizwana chaudhri, Holy family hospital, Rawalpindi, Pakistan, The study was published in journal of Rawalpindi medical college and concluded that rectal diclofenac should be further promoted , for pain relief, in women following episiotomy.

ELIGIBILITY:
Inclusion Criteria:

1. age: 20:35 years.
2. Primigravidae as elective procedure.
3. face to pubis delivery.
4. Big baby.
5. Narrow pelvic arch.
6. Elderly primigravida.
7. old perineal scar as episiotomy or perineorrhaphy.
8. Manipulative delivery.
9. To cut short second stage cases such as pre eclampsia.
10. Premature baby.
11. Fetal distress.

Exclusion Criteria:

1. more than 35 years.
2. pelvic inflammatory disease.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1024 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Post episiotomy pain relief | First three days after delivery
  The relief of pain after delivery measured by pain relief scale..Pain relief scale Title: pain intensity scale Minimum 0 means no pain Maximum 4 means severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Diaa eldin Mohammed, Professor, Study Chair — women health hospital assiut university; Osama Saber, Lecturer, Study Director — women health hospital assiut university

IPD SHARING:
Plan to Share IPD: Yes
Iidentify individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be available for sharing within 6 month of completion of the study
Access Criteria: Data access requests will be reviewed by an external independent review panel.requestorswill be required to sign a data access agreement
URL: http://www.aun.edu.eg

REFERENCES:
- See also: Worldwide website written collaporatively by people who use it — https://en.m.wikipedia.org/wiki/Episiotomy
- See also: a free search engine accessing primarily the MEDLINE database of references and abstracts on life sciences and biomedical topics — https://pubmed.ncbi.nlm.nih.gov/17465071